CLINICAL TRIAL: NCT07330518
Title: Comparison of Conventional Buccal Nerve Block Versus Buccal Nerve Trunk Block for Anaesthesia of Buccal Mucosa During Extraction of Mandibular Posterior Teeth
Brief Title: Comparison of Conventional Buccal Nerve Block Versus Buccal Nerve Trunk Block During Extraction of Posterior Mandibular Teeth
Acronym: Buccal Trunk
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Watim Medical & Dental College (Other)
Responsible Party: Principal Investigator, SYED SAAD AFTAB, Principal Investigator, Watim Medical & Dental College
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: WM&DCR/R&D(ERB)/2023/68
Record Dates: First submitted 2025-12-08; First posted 2026-01-09 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2025-12

CONDITIONS: Pain (Visceral, Somatic, or Neuropathic)
Keywords: Buccal Trunk Block
MeSH Terms: conditions — Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Conventional Buccal Nerve Block for anesthesia of buccal mucosa (Experimental): Administration of anesthesia using conventional buccal nerve block technique for anesthesia of buccal mucosa.
  Interventions: Procedure: Conventional Buccal Nerve Block
- Buccal Nerve Trunk Block (Experimental): Administration of anesthesia at the buccal trunk 10mm above the coventional buccal nerve block for anesthesia of buccal mucosa.
  Interventions: Procedure: Buccal Nerve Trunk Block

INTERVENTIONS:
Procedure: Conventional Buccal Nerve Block — Arm Description: Administration of anesthesia at the level of occlusion lateral to last mandibular molar. Needle is inserted until bone contact is achieved. 1ml lidocaine with 1:100000 anesthesia is administered.
  Arms: Conventional Buccal Nerve Block for anesthesia of buccal mucosa
Procedure: Buccal Nerve Trunk Block — Arm Description: Administration of anesthesia 10 mm above occlusal plane lateral to last mandibular molar. 1ml lidocaine with 1:100000 anesthesia is administered.
  Arms: Buccal Nerve Trunk Block

SUMMARY:
This randomised control trial will compare the efficacy of conventional buccal nerve block versus buccal trunk block using visual analogue scale to evaluate pain and additional anesthesia injection during extraction of mandibular molars.

DETAILED DESCRIPTION:
Dental extraction of mandibular posterior teeth require buccal mucosa anesthesia for pain free extraction. Conventional buccal nerve block is the commonly used technique for anesthesia of buccal mucosa but often is not effective and requires multiple injections. This study aims to compare coventional buccal nerve block with buccal nerve trunk block on the basis of Efficacy of local anesthesia which will be determined by need for supplemental infiltration: Use of more than 1 anesthesia cartridges during procedure will be labelled as need for supplemental infiltration.

Intraoperative pain perception: It was assessed while giving injection and during extraction of the tooth using the visual analog scale (VAS) scores. Score of more than 4 will be labelled as positive pain perception.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 20 to 60 years
* Patients of both gender
* Patient requiring extraction of mandibular molars

Exclusion Criteria:

* Pregnant women
* Pathologies associated with teeth i.e. cysts, tumors
* Patients on radiotherapy or chemotherapy
* Patients with mandibular fracture

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 100 (Estimated)
Dates: Start 2026-03-20 (Estimated); Primary Completion 2027-01-01 (Estimated); Study Completion 2027-01-01 (Estimated)

PRIMARY OUTCOMES:
Intraoperative pain perception | Within 2hours of anesthesia administration
  It was assessed while giving injection and during extraction of the tooth using the visual analog scale (VAS) scores. Facial pain scale uses facial expression to evaluate the amount of pain. It has scores ranging from 0 to 10 with 0 as the least pain and 10 as the worst pain. Score of more than 4 will be labelled as positive pain perception.
Need for supplemental infiltration | Within 2 hour of initial anesthesia administration
  Use of more than 1 anesthesia cartridges during procedure will be labelled as need for supplemental infiltration.

CONTACTS AND LOCATIONS:
Locations (1):
- Watim Medical College & Dental Hospital, Islamabad, Islamabad, Pakistan, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] 1.Risbaf-Fakoor S, Hashemzehi H, Jahantigh H, Arab K, Gholami L. Adjunctive low-level laser therapy using 980-nm diode laser after impacted mandibular third molar surgery: a randomized clinical trial. Avicenna J Clin Med. 2020; 26 (4):199-205. 2.Mahat A, Yadav R, Yadav A, Acharya P, Dongol A, Sagtani A et al. A comparative study of the effect of sutureless versus multiple sutures technique on complications following third molar surgery in Nepalese subpopulation. Int J Dent. 2020; 2020(1):1-6. 3.Sruthi MA, Ramakrishnan M. Transpapillary injection technique as a substitute for palatal infiltration: a split-mouth randomized clinical trial. Int J Clin Pediatr Dent. 2021; 14(5):640-3. 4.Decloux D, Ouanounou A. Local anaesthesia in dentistry: a review. Int Dent J. 2020; 71(2):87-95. 5.Wang YH, Wang DR, Liu JY, Pan J. Local anesthesia in oral and maxillofacial surgery: A review of current opinion. J Dent Sci. 2021; 16(4):1055-65. 6.Koyata T, Yanai C, Shionoya Y, Takasugi Y, Sunada K. Buccal nerve trunk block anesthetizes the buccal mucosa beyond the papilla of the parotid duct. J Oral Maxillofac Surg. 2023;81(3):272-9. 7.Figueiredo R, Sofos S, Soriano-Pons E, Camps-Font O, Sanmarti-Garcia G, Gay-Escoda C, Valmaseda-Castellón E. Is it possible to extract lower third molars with infiltration anaesthesia techniques using articaine? A double-blind randomized clinical trial. Acta Odontol. Scand. 2021 Jan 2;79(1):1-8.